CLINICAL TRIAL: NCT07059416
Title: The Effect of Mindful Hand Hygiene Practice on Self-Care Perception and Self-Compassion Levels of Oncology Nurses; Mixed Design Example
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024028
Record Dates: First submitted 2025-05-11; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Mindfulness Meditation; Selfcompassion
Keywords: oncology nursing, mindfulness, self-compassion, self-care
MeSH Terms: interventions — Hand Sanitizers

STUDY DESIGN:
Intervention Model Description: In this context, the prototype model of the pretest-posttest control group design is presented as follows:
  R-Randomization Experimental Group T1-Pretest G-Intervention T2-Posttest Control Group T1-Pretest T2-Posttest. Before the pre-intervention groups were assigned, the first tests were applied, hand hygiene practice was taught with conscious awareness and they were asked to apply the hand hygiene ritual while performing the hand hygiene steps for four weeks. Four weeks after the beginning of the study, data were collected again with data collection tools.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): Oncology nurses practice mindfulness hand hygiene for four weeks
  Interventions: Behavioral: Oncology nurses carried out hand hygiene awareness activities with positive affirmation words and breathing exercises while washing hands or providing hand hygiene with hand antiseptic.
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Oncology nurses carried out hand hygiene awareness activities with positive affirmation words and breathing exercises while washing hands or providing hand hygiene with hand antiseptic. — positive affirmation, focus on the moment
  Arms: İntervention group

SUMMARY:
This study was planned to evaluate the effect of hand hygiene awareness activities to be carried out by nurses with positive affirmation words and breathing exercises during hand washing or hand hygiene with hand antiseptic on increasing the conscious awareness and self-compassion of oncology nurses and to determine the experiences of oncology nurses regarding hand hygiene awareness activities.

Research Hypothesis Hypothesis 1a: Hand hygiene with awareness increases the conscious awareness levels of oncology nurses.

Hypothesis 1b: Hand hygiene with awareness increases the self-compassion levels of oncology nurses.

Hypothesis 1c: Hand hygiene with awareness increases the self-care perception levels of oncology nurses.

Research Question: How does hand hygiene with awareness affect the self-compassion, self-care perception and conscious awareness levels of oncology nurses?

DETAILED DESCRIPTION:
This study was planned according to the nested mixed design method in order to test the effect of the awareness hand hygiene practice applied by oncology nurses working in the bone marrow transplantation unit and hematological oncology clinic on the self-compassion, self-care perception and conscious awareness levels of the nurses and to obtain in-depth predictions. This study was conducted with oncology nurses working in the oncology clinics of a university hospital in Ankara between 10.01.2025-10.04.2025. A randomized controlled design was used to collect the quantitative data of the study. The basic feature of the pre-test-post-test control group design was to randomly assign the subjects to both groups in order to control the variables that may have an effect on the outcome variable. The universe of the study will consist of the nurses of the bone marrow transplantation unit and hematological oncology clinic where the study will be conducted. G*Power 3.1.9.7 program was used to calculate the sample size. This study was conducted with a total of 44 nurses, 23 in the intervention group and 21 in the control group. Inclusion criteria will be nurses who have been working as oncology nurses for at least one year and volunteered to participate in the study.

Exclusion Criteria of the Study: Having done/having done regular activities related to mindfulness or self-compassion such as meditation, yoga, etc. in the last year.

Randomization: Nurses who met the inclusion criteria were randomly and equally divided into 2 groups as the experimental group and the control group using a computer-based program (www.random.org). The assignment to the experimental and control groups will be made by an independent statistician in order to ensure confidentiality and prevent bias. The data was coded as 'A' and 'B' by the researcher and transferred to the computer. In addition, the analysis of the coded data was performed by an independent statistician in order to prevent bias in the evaluation of the data. After the consents of the patients who met the inclusion criteria were obtained and the pre-tests were completed, they were assigned to the groups according to the assignment list.

Blinding: Due to the nature of the study, blinding will not be applied to the participants. The statistical analysis of the data was performed by an independent statistician who did not know the groups. In this way, bias will be prevented during the data analysis stage.

Data Collection Before Assignment to Groups: Information about the research will be provided, and the compliance of the nurses who agree to participate in the research with the inclusion criteria will be assessed. After the written consent of the nurses who meet the inclusion criteria is obtained, the nurses will be invited to fill out the Personal Information Form, Watson Healing Self-Assessment Scale, Conscious Awareness Scale and Self-Compassion Scale-Short Form. The sealed envelope where the randomization was made will be opened and the nurse will be assigned to the experimental or control group.

Intervention Group: A three-hour training on conscious awareness will be given to the nurses assigned to the intervention group. Information will be provided on the "Hand Hygiene Practice with Awareness" practice and a hand hygiene awareness practice will be carried out together. The researcher will check whether the nurse has implemented the hand hygiene awareness practice correctly during this process. The nurse will be asked to do this hand hygiene awareness while passing from one patient to another for eight weeks. In order to increase compliance with the hand hygiene awareness application, the researcher will give the nurses an exercise record form and send them a daily message to remind them of the hand hygiene awareness application. The messages will be used to check whether the nurse has any problems with the exercise. At the end of the fourth week, the participants will be invited to fill out the Watson Healing Self-Assessment Scale, Watson Healing Self-Assessment Scale, Conscious Awareness Scale and Self-Compassion Scale-Short Form.

ELIGIBILITY:
Inclusion Criteria: and volunteering to participate in research

* Having worked as an oncology nurse for at least one year
* Volunteering to participate in research

Exclusion Criteria:

* Having done/having done regular activities such as meditation, yoga, etc. related to mindfulness or self-compassion in the last year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
1. oncology nurses' conscious awareness levels 2. oncology nurses' self-compassion levels 3. oncology nurses' self-care perception levels | four weeks
  The Watson Caritas Self-Rating Score for oncology nurses' self-care perception levels Short Form of the Self-Compassion Scale for oncology nurses' self-compassion levels Mindful Attention Awareness Scale for oncology nurses' conscious awareness levels

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay University, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol including conscious hand hygiene practice
Supporting Information: Study Protocol